CLINICAL TRIAL: NCT01003990
Title: Atazanavir (BMS-232632) for HIV Infected Individuals Completing Atazanavir Clinical Trials: An Extended Access Study
Brief Title: Roll-Over Protocol To Provide Atv And/Or Truvada For Extended Access
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AI424-077
Record Dates: First submitted 2009-10-20; First posted 2009-10-29 (Estimated); Results first posted 2017-05-11 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-04

CONDITIONS: HIV
Keywords: Treatment experienced
MeSH Terms: interventions — Atazanavir Sulfate; atazanavir, ritonavir drug combination; Tenofovir; Emtricitabine; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Lopinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Atazanavir (Experimental)
  Interventions: Drug: Atazanavir
- Atazanavir/Ritonavir (Experimental)
  Interventions: Drug: Atazanavir/Ritonavir
- Lopinavir/Ritonavir (Active Comparator): Ritonavir-boosted Lopinavir (LPV/RTV 400/100 mg) administered twice a day (BID) with Tenofovir/ Emtricitabine (TDF/FTC).
  Interventions: Drug: Tenofovir/Emtricitabine; Drug: Lopinavir/ritonavir

INTERVENTIONS:
Drug: Atazanavir — Tablets, Oral, 400 mg, once daily, indefinitely
  Other Names: Reyataz; BMS-232632
  Arms: Atazanavir
Drug: Atazanavir/Ritonavir — Tablets, Oral, 300/100 mg, once daily, indefinitely
  Other Names: Reyataz; BMS-232632
  Arms: Atazanavir/Ritonavir
Drug: Tenofovir/Emtricitabine — Tablets, Oral, 300/200 mg, once daily, indefinitely
  Other Names: Truvada
  Arms: Lopinavir/Ritonavir
Drug: Lopinavir/ritonavir — Tablets, Oral, 400/100 mg, twice daily, indefinitely
  Arms: Lopinavir/Ritonavir

SUMMARY:
The purpose of this study is to provide atazanavir or tenofovir-emtricitabine to HIV-infected subjects who have completed atazanavir or tenofovir-emtricitabine therapy on a previous BMS sponsored clinical trial and to collect long-term safety information on the treated population.

DETAILED DESCRIPTION:
Provide study drug for patients rolling off BMS ATV clinical trials in countries where these medications are not commercially available.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must provide written informed consent
* Currently receiving atazanavir (unboosted or boosted with 100 mg ritonavir QD)and/or tenofovir-emtricitabine at time of screening and viral load is

  ≤ 10,000 copies/mL while on therapy
* Subjects who are receiving investigational antiretroviral agents through Expanded Access Programs will be allowed to participate following discussion and approval by the BMS Medical Monitor
* ≥ 16 years of age (or minimum age as determined by local regulatory or as legal requirements dictate)
* Both females of child-bearing potential and males must utilize effective barrier contraception to reduce transmission of sexually transmitted diseases, including HIV. Other contraception in addition to barrier methods are permitted, however interactions between atazanavir and oral contraceptives have not been studied

Exclusion Criteria:

* WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 8 weeks after the study
* WOCBP using a prohibited contraceptive method (no contraceptive methods prohibited in this study. However, caution is warranted with coadministration of oral contraceptives)
* Women who are pregnant or breastfeeding
* Women with a positive pregnancy test on enrollment or prior to study drug administration, with the exception of women rolling over from AI424182, who may still have a positive β-HCG test at the time of enrollment
* All subjects previously discontinued from an atazanavir study for any reason
* Active alcohol or substance abuse sufficient, in the Investigator's opinion, to prevent adequate compliance with study therapy or to increase the risk of developing pancreatitis or chemical hepatitis
* Any other clinical conditions or prior therapy that, in the opinion of the investigator, would make the subject unsuitable for study, or unable to comply with the dosing requirements
* Any of the following laboratory values:
* a) Serum creatinine ≥ 1.5 times the upper limit of normal,
* b) Liver enzymes (AST, ALT) ≥ 5 times the upper limit of normal,
* Hypersensitivity to any component of the formulation of study drug
* Refer to Section 6.4.1 which details all prohibited therapies
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious disease) illness must not be enrolled into this study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 710 (Actual)
Dates: Start 2002-10; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (68):
- United States (12):
  - Phoenix Body Positive, Inc, Phoenix, Arizona
  - Rand Schrader Clinic, Los Angeles, California
  - St Francis Memorial Hospital, San Francisco, California
  - Sbma Research, Llc, Miami Beach, Florida
  - St Josephs Cmprhnsv Rsch Inst, Tampa, Florida
  - Infectious Disease Of Indiana, Psc, Indianapolis, Indiana
  - Univ Of Kansas Sch Of Med, Wichita, Kansas
  - Cri Of New England, Boston, Massachusetts
  - University Of Nebraska Medical Center, Omaha, Nebraska
  - Jemsek Clinic, Huntersville, North Carolina
  - Tarrant County Inf Dis Assoc, Fort Worth, Texas
  - The Schrader Clinic, Houston, Texas
- Argentina (3):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Córdoba, Córdoba Province
  - Local Institution, Rosario, Santa Fe Province
- Brazil (7):
  - Local Institution, Curitiba, Paraná
  - Local Institution, Recife, Pernambuco
  - Local Institution, Rio de Janeiro, Rio de Janeiro
  - Local Institution, Rio de Janeiro - Rj, Rio de Janeiro
  - Local Institution, Campinas, São Paulo
  - Local Institution, Sao Paulo - Sp, São Paulo
  - Local Institution, São Paulo, São Paulo
- Canada (2):
  - Local Institution, Hamilton, Ontario
  - Local Institution, Montreal, Quebec
- Local Institution, Santiago, Santiago Metropolitan, Chile
- Local Institution, Bogota, Cundinamarca, Colombia
- Local Institution, San José, Barrio Aranjuez, Costa Rica
- Local Institution, Santo Domingo, Dominican Republic
- France (4):
  - Local Institution, Le Kremlin-Bicêtre
  - Local Institution, Lyon
  - Local Institution, Paris
  - Local Institution, Tourcoing
- Local Institution, Guatemala City, Guatemala
- Local Institution, Budapest, Hungary
- Local Institution, Jakarta, Indonesia
- Italy (4):
  - Local Institution, Milan
  - Local Institution, Modena
  - Local Institution, Roma
  - Local Institution, Torino
- Local Institution, Kuala Lumpur, Kuala Lumpur, Malaysia
- Local Institution, Mexico City, Mexico City, Mexico
- Local Institution, Panama City, Panama
- Peru (2):
  - Local Institution, Lima, Lima Province
  - Local Institution, Barranco, Lima region
- Portugal (2):
  - Local Institution, Lisbon
  - Local Institution, Porto
- Puerto Rico (2):
  - Clinical Research Puerto Rico, Inc., San Juan
  - V.A. Medical Center, San Juan
- Russia (2):
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
- Local Institution, Singapore, Singapore
- South Africa (7):
  - Local Institution, Port Elizabeth, Eastern Cape
  - Local Institution, Bloemfontein, Free State
  - Local Institution, Johannesburg, Gauteng
  - Local Institution, Meadowdale, Gauteng
  - Local Institution, Westdene, Gauteng
  - Local Institution, Observatory, Western Cape
  - Local Institution, Rugby, Western Cape
- Spain (6):
  - Local Institution, Badalona
  - Local Institution, Barcelona
  - Local Institution, Bilbao
  - Local Institution, Córdoba
  - Local Institution, Madrid
  - Local Institution, Seville
- Taiwan (2):
  - Local Institution, Kaohsiung City
  - Local Institution, Taipei
- Thailand (2):
  - Local Institution, Bangkok
  - Local Institution, Chiang Mai

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 710 participants were enrolled, 709 were treated. The participant who did not receive treatment was enrolled in error having been assigned to efavirenz in the parent study AI424034 (only subjects assigned to ATV rolled over into AI424077).
Groups:
- Atazanavir (ATV): Atazanavir: Tablets, Oral, 400 mg (2 x 200 mg capsules), once daily with food, indefinitely
- Atazanavir/Ritonavir (ATV/RTV): Ritonavir-boosted Atazanavir (ATV/RTV 300/100 mg). Tablets administered orally once daily (QD) with food, indefinitely.
  Ritonavir: 100 mg QD Atazanavir: 300 mg QD (3 x 100 mg capsules, or 2 x 150 mg capsules)
- Lopinavir/Ritonavir (LPV/RTV): Ritonavir-boosted Lopinavir (LPV/RTV 400/100 mg) administered twice a day (BID) with Tenofovir/ Emtricitabine (TDF/FTC).
  Lopinavir: 400 mg BID Ritonavir: 100 mg BID Tenofovir/Emtricitabine: Tablets, Oral, 300/200 mg, once daily (QD) with food, indefinitely (one tablet with 300 mg - 200 mg QD)
Period: Overall Study
Arm/Group | Atazanavir (ATV) | Atazanavir/Ritonavir (ATV/RTV) | Lopinavir/Ritonavir (LPV/RTV)
Started | 459 | 154 | 96
Completed | 367 | 103 | 53
Not Completed | 92 | 51 | 43
Not completed — Adverse Event | 8 | 5 | 11
Not completed — Death | 0 | 8 | 1
Not completed — Lack of Efficacy | 10 | 2 | 3
Not completed — Lost to Follow-up | 30 | 12 | 7
Not completed — Reasons Not Identified | 14 | 13 | 8
Not completed — Poor/Non-compliance | 4 | 3 | 2
Not completed — Pregnancy | 10 | 2 | 4
Not completed — No Longer Met Study Criteria | 4 | 1 | 0
Not completed — Subject Withdrew Consent | 12 | 5 | 7

BASELINE CHARACTERISTICS:
Population: All Treated Participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Atazanavir (ATV) | Atazanavir/Ritonavir (ATV/RTV) | Lopinavir/Ritonavir (LPV/RTV) | Total
Number analyzed (Participants) | 459 | 154 | 96 | 709
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.6 (9.00) | 35.9 (8.81) | 37.6 (10.16) | 36.6 (9.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 172 | 54 | 30 | 256
  Male | 287 | 100 | 66 | 453
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 158 | 34 | 18 | 210
  Black or African American | 112 | 25 | 2 | 139
  American Indian/Alaska Native | 1 | 0 | 0 | 1
  Asian | 53 | 13 | 18 | 84
  Other | 135 | 82 | 58 | 275

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs), Treatment Related SAEs, Treatment Related Adverse Events (AEs), AEs Leading to Discontinuation of Study Therapy, Grade 3 to Grade 4 AEs, Grade 3 to Grade 4 AEs, CDC Class C AIDS Events, or Death
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=having certain, probable, possible, or missing relationship to study drug. Grade (Gr) 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4= Potentially Life-threatening or disabling. AIDS Defining Diagnosis ( CDC Class C AIDS Events) are identified from HIV Related Diagnosis.
Time Frame: Date of First Dose to 30 days post the last dose; approximately 405 weeks)
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Atazanavir (ATV) | Atazanavir/Ritonavir (ATV/RTV) | Lopinavir/Ritonavir (LPV/RTV)
Number analyzed (Participants) | 459 | 154 | 96
Participants
  SAEs | 35 | 19 | 12
  Treatment Related SAEs | 4 | 1 | 0
  Treatment Related AEs of Any Grade | 180 | 49 | 34
  AEs Leading to Discontinuation of Study Therapy | 8 | 5 | 11
  Grade 3 to Grade 4 AEs | 72 | 27 | 15
  Grade 2 to Grade 4 AEs | 102 | 28 | 19
  CDC Class C AIDS Events | 2 | 0 | 0
  Deaths | 2 | 7 | 1

ADVERSE EVENTS:
Time Frame: Date of first dose to date of last dose plus 30 days; approx. 680 weeks
Description: All Treated Participants
  Study Initiated: November 13, 2002 Study Completion: February 16, 2016
Groups:
- Atazanavir/Ritonavir (ATV/RTV): Ritonavir-boosted Atazanavir (ATV/RTV 300/100 mg). Tablets administered orally once daily (QD) with food, indefinitely.
  Ritonavir: 100 mg QD; Atazanavir: 300 mg QD (3 x 100 mg capsules, or 2 x 150 mg capsules)
- Lopinavir/Ritonavir (LPV/RTV): Ritonavir-boosted Lopinavir (LPV/RTV 400/100 mg) administered twice a day (BID) with Tenofovir/ Emtricitabine (TDF/FTC).
  Lopinavir: 400 mg BID; Ritonavir: 100 mg BID; Tenofovir/Emtricitabine: Tablets, Oral, 300/200 mg, once daily (QD) with food, indefinitely (one tablet with 300 mg - 200 mg QD)
Arm/Group | Atazanavir (ATV) | Atazanavir/Ritonavir (ATV/RTV) | Lopinavir/Ritonavir (LPV/RTV)
All-Cause Mortality (participants affected / at risk) | 2/459 | 7/154 | 1/96
Serious Adverse Events (participants affected / at risk) | 35/459 | 19/154 | 12/96
Other Adverse Events (participants affected / at risk) | 284/459 | 92/154 | 57/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atazanavir (ATV) (N=459) | Atazanavir/Ritonavir (ATV/RTV) (N=154) | Lopinavir/Ritonavir (LPV/RTV) (N=96)
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Accidental exposure to product (Injury, poisoning and procedural complications) | 0 | 1 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Cervicitis (Infections and infestations) | 0 | 1 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 2 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Leukaemoid reaction (Blood and lymphatic system disorders) | 0 | 1 | 0
Major depression (Psychiatric disorders) | 2 | 0 | 0
Neurosyphilis (Infections and infestations) | 0 | 0 | 1
Open fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0 | 1
Abdominal infection (Infections and infestations) | 0 | 1 | 0
Proctitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0 | 0
Uterine disorder (Reproductive system and breast disorders) | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 1
Abortion (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 0
Appendiceal abscess (Infections and infestations) | 1 | 0 | 0
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Hepatitis A (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 2 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0 | 0
Traumatic ulcer (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tuberculosis (Infections and infestations) | 0 | 1 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 1 | 0
Bicytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Gallbladder polyp (Hepatobiliary disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 1 | 0
Oedema (General disorders) | 0 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Acute abdomen (Gastrointestinal disorders) | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0
Acute psychosis (Psychiatric disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 0
Gastric ulcer perforation (Gastrointestinal disorders) | 1 | 0 | 0
Hodgkin's disease nodular sclerosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Infective tenosynovitis (Infections and infestations) | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0
Testicular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 1 | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1 | 1
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Extrapulmonary tuberculosis (Infections and infestations) | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 | 0 | 0
Endometrial hypertrophy (Reproductive system and breast disorders) | 0 | 1 | 0
Mastoiditis (Infections and infestations) | 0 | 0 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Atazanavir (ATV) (N=459) | Atazanavir/Ritonavir (ATV/RTV) (N=154) | Lopinavir/Ritonavir (LPV/RTV) (N=96)
Alanine aminotransferase increased (Investigations) | 27 | 5 | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 45 | 3 | 1
Nasopharyngitis (Infections and infestations) | 51 | 32 | 24
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 7 | 6
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 6 | 7 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 27 | 13 | 12
Diarrhoea (Gastrointestinal disorders) | 47 | 22 | 12
Urinary tract infection (Infections and infestations) | 11 | 11 | 2
Abdominal pain upper (Gastrointestinal disorders) | 13 | 2 | 6
Influenza (Infections and infestations) | 32 | 16 | 6
Abdominal pain (Gastrointestinal disorders) | 20 | 8 | 4
Creatinine renal clearance decreased (Investigations) | 0 | 16 | 8
Headache (Nervous system disorders) | 37 | 15 | 8
Jaundice (Hepatobiliary disorders) | 24 | 5 | 1
Upper respiratory tract infection (Infections and infestations) | 74 | 10 | 4
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 6
Blood bilirubin increased (Investigations) | 34 | 3 | 1
Bronchitis (Infections and infestations) | 32 | 8 | 6
Gastritis (Gastrointestinal disorders) | 12 | 8 | 3
Nausea (Gastrointestinal disorders) | 19 | 4 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 | 12 | 5
Blood cholesterol increased (Investigations) | 0 | 4 | 7
Ocular icterus (Eye disorders) | 31 | 4 | 0
Pyrexia (General disorders) | 12 | 9 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.